CLINICAL TRIAL: NCT03132753
Title: Developing SUPPORT, a Community-Driven, Recovery-Oriented System of Care
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michelle Salyers, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1511731907
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUPPORT Group (Experimental): Subjects enrolled in the intervention.
  Interventions: Behavioral: SUPPORT
- Treatment as Usual (No Intervention): Subjects enrolled in standard services.

INTERVENTIONS:
Behavioral: SUPPORT — SUPPORT clients will be offered 12 months of support service with a recovery coach. The recovery coach will guide the client through their recovery, offering guidance and support, while coordinating their treatment services, including support services. The program will provide clients with up to $700 worth of vouchers to cover the cost of additional flexible support services over the 12 months of program enrollment, which will be personalized to fit the needs of the client. These cost vouchers will cover support services, such as housing, employment services, substance use treatment, transportation, childcare, educational or vocational services, or aftercare planning. The costs of each service is determined by the service provider. Further, the recovery coach will assist the client in choosing appropriate services and coordinating/monitoring service completion.
  Arms: SUPPORT Group

SUMMARY:
The investigators seek to develop and assess the effectiveness of Substance Use Programming for Person-Oriented Recovery and Treatment (SUPPORT), a community-driven recovery-oriented system of care for individuals recently released from prison. SUPPORT is modeled after Indiana Access to Recovery (ATR), a program that operated between October 2007 and December 2014. ATR, a national initiative funded by the Substance Abuse and Mental Health Services Administration (SAMHSA), provided comprehensive, flexible, recovery-oriented services for substance use disorder (SUD). The investigators' local evaluation of this program demonstrated significant improvement in a number of recovery-related outcomes (e.g., substance use, employment, income, involvement in the criminal justice system, and emotional well-being) for clients between intake and discharge. Additionally, qualitative findings from this evaluation demonstrated ATR was well liked among clients and providers. While Indiana ATR did serve a wider range of clients, the investigators have focused SUPPORT on returning inmates because (a) this was the largest group served by the program and (b) there is significant need for evidence-based SUD interventions for this population.

The investigators' primary long-term goal is to establish an effective and scalable recovery-oriented system of care for SUD within the reentry population. The investigators will conduct a pilot test comparing SUPPORT clients to clients receiving usual treatment. The investigators will collect quantitative data for both groups at multiple time points to understand the intervention's impact on recovery capital and outcomes and will collect qualitative data from SUPPORT clients to better understand their program and post-discharge experiences.

DETAILED DESCRIPTION:
The investigators will conduct the pilot at Public Advocates in Community Re-Entry (PACE), a nonprofit that provides services to individuals with felony convictions in Marion County Indiana. PACE has provided re-entry services in Marion County, IN for 55 years. PACE's services are divided into four distinct categories: transitional, employment, addiction, and pre-release services. It is the only former ATR agency in Marion County specializing in a re-entry population, and our evaluation of Indiana's program demonstrated they had significantly lower rates of recidivism than any other Marion County agency. In 2015, PACE served 1,703 new clients.

The investigators will recruit 100 clients for participation in the pilot, half (50) will be assigned to SUPPORT and half (50) to treatment as usual. SUPPORT clients will be offered 12 months of support service with a PACE recovery coach. The recovery coach will guide the SUPPORT client through their recovery, offering guidance and support, while coordinating their treatment services, including support services. The SUPPORT program will provide SUPPORT clients with $1,000 worth of vouchers to cover the cost of additional flexible support services over the 12 months of program enrollment, which will be personalized to fit the needs of the client. These cost vouchers will cover similar support services as the previous Access to Recovery (ATR) program, such as housing (permanent, transitional), employment services (training, placement, readiness), substance use treatment, transportation, childcare, educational or vocational services, or aftercare planning. The costs of each service is determined by the service provider. Clients will NOT be responsible for keeping track of their vouchers, but rather, his/her assigned recovery coach will track all voucher funding/spending. Further, the recovery coach will assist the client in choosing appropriate services and coordinating/monitoring service completion.

Clients in the treatment as usual group will have significantly reduced choices in services compared to SUPPORT clients. These clients will not receive vouchers to access support services such as transportation and housing and will only receive standard case management, which is more prescriptive and less intensive than the recovery consultant services provided through SUPPORT.

All PACE clients who are over the age of 18, have a SUD, are no longer incarcerated (in a prison, jail, or work release facility), are within 3 months from their release from prison, jail, or work release, and are unable to access the previously mentioned Recovery Works program, will be eligible for study participation. For both parolees and probationers the risk of recidivism is highest in the first year of release; therefore, the investigators will be connecting with clients during the initial months following releases. The investigators will also be excluding sex offenders from the pilot, as they face greater barriers to community integration and experience higher levels of supervision while on parole, which have the potential to confound results during a small-scale pilot. Once a potential client is released from incarceration and enrolled at PACE, if eligible, an intake worker will inform them of the opportunity to participate in the pilot study and describe the SUPPORT program services. If the client agrees to participate in the pilot, they will sign a consent form and be randomly assigned to either SUPPORT or a treatment as usual condition. If a participant in either the SUPPORT or treatment as usual group is re-incarcerated during the study period, the investigators will not engage them while under correctional supervision to collect data and the investigators will replace them with a new participant. However, if a participant is re-incarcerated but released back into the community during the study period, and reengages with PACE, they will continue to be a part of the study and the investigators will continue to collect data and offer them SUPPORT services. In short, for the purposes of this pilot, the investigators will not be collecting data from clients while incarcerated.

Quantitative:

PACE will hire and assign two recovery coaches to provide SUPPORT services for the pilot. Once hired, the recovery coaches will complete all required IRB training and receive training on data collection and the informed consent procedures. The names of these recovery coaches will be added to the IRB protocol through an IRB amendment, having completed all required training, before interacting with subjects.

In addition to providing the support services, recovery coaches will 1) go over the statement of informed consent and Authorization form and have willing participants provide their signature, 2) conduct an initial interview with all clients after they have provided informed consent (to be included at the beginning of the electronic data collection) and have been assigned to the SUPPORT or comparison group, and 3) collect electronic data using REDCap system at the designated time points. Recovery consultants will collect data through a computer assisted personal interview (CAPI) (i.e., individual interviews assisted by computer technology.) Consultants will conduct interviews in a private room, away from other individuals so that others may not overhear what is discussed. Each consultant will have a tablet computer through which they will access the REDCap system. After the consultant has collected all necessary service or background data, the REDCap system will instruct them to hand the tablet over to the client to allow them to answer the remaining questions (regarding Self Determination, Treatment Motivation, Self Efficacy, Stages of Change, Substance Use, and Quality of Life) independently. The recovery coach will hand the tablet to the client and move so they cannot see their responses. Instructions will appear on the tablet telling the client to ask questions should they need assistance with either the tablet or answering a question. Should the client need assistance using the tablet or answering a question, the recovery coach will be available to help. During the screening process (i.e. client enrollment), client illiteracy will be picked up. Should a client be illiterate, they will still be invited to participate, but a recovery coach will read the questions rather than asking them to answer the questions independently.

CAPI interviews will be conducted with all clients (SUPPORT and non-SUPPORT) at baseline and 6 and 12 months to understand change in outcomes overtime. Consultants will also conduct a CAPI interview at 15 months with SUPPORT clients only to understand retention of treatment effects three months post discharge. Based on our previous experience conducting CAPI interviews, the investigators expect this process to take between 60 and 90 minutes.

CAPI Data collection measures include: demographic and background information on all clients at baseline; including: date of birth, gender, race, ethnicity, sexual orientation, housing history, education, employment history, and past involvement in addiction recovery and treatment. The investigators will also collect a number of measures, including (1) agency/self-determination, (2) recovery capital (i.e. treatment motivation, social support/networks, and self-efficacy), and (3) recovery-related outcomes (frequency of substance use and abstinence, incremental progress towards recovery, quality of life, recidivism, and administrative data on housing status, education, employment, income, physical and mental health status, and attendance at self-report self-help groups.)

Additionally, IU researchers will conduct structured social network interviews within one week of the client's entrance in the study and at 12 months. Social support is a proven influential factor on recovery. Having relationships and social networks that provide support, friendship, love, and hope through the process of recovery improves outcomes. The recovery coaches that work in the SUPPORT program will work with the clients to utilize their recovery support services to strengthen the individual's place in the community as a productive community member, family member, and worker, and, ideally, improve the quality of clients' interpersonal relationships and likelihood of positive recovery outcomes. This study will measure social support as a recovery-related outcome to see if the program is able to positively impact the social support in clients' lives over the course of 12 months. The total data collection time for these interviews will be between 30 and 60 minutes depending on the number of individuals in the client's network. At the time of the second network interview, the investigators will also collect qualitative data on SUPPORT client's overall program experience. During these interviews, the client will be asked for the first names and last initial of people who provide certain types of social support in his/her life.

Qualitative:

IU researchers will also collect qualitative data from both group through semi-structured interviews. The purpose of the interviews is to develop an understanding of client's treatment experience and how the SUPPORT program may have assisted them in overcoming barriers to recovery. These interviews are expected to take between 45 and 60 minutes. Guiding questions for the interview include: "Describe what you liked/did not like about the SUPPORT program (probe: client-centeredness, self-determination)."; "How was your relationship with your recover consultant?"; "Overall, how has the program helped you in your recovery? (probe: motivation; social capital; quality of life; elimination of barriers)"; "Are there specific things the program helped you with that you would not have been able to do on your own?"; "How did the program help you not return to jail (for those who did not recidivate)/How could the program have assisted your better so you would not have returned to jail (for those who did recidivate)?"; "If you experienced a relapse in the program, how did the program help you through that?"; "If you could change anything about SUPPORT, what would it be? Why?" (Attachment: Qualitative Interview Questions)

Also, researchers will conduct focus groups with SUPPORT clients after their 15-month CAPI interview. The researchers will conduct between 5 and 8 focus groups with 5-10 participants each. The researchers will attempt to recruit all SUPPORT clients for focus groups. Focus groups will last between 60 and 90 minutes and will be audio recorded.

ELIGIBILITY:
Inclusion Criteria:

* All PACE clients who are over the age of 18, have a SUD, are no longer incarcerated (in a prison, jail, or work release facility), are within 3 months of release from prison, jail, or work release, and are unable to access the previously mentioned Recovery Works program will be eligible for study participation.

Exclusion Criteria:

* Any individual that is not a PACE client, has not been released from prison, over the age of 18, or does not have a substance abuse disorder will not be included in the study.

Also, sex offenders will be excluded from this study because of the additional integration barriers faced by this population and their increased parole supervision, as these may confounding variables in such a small pilot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Advocates in Community Re-Entry (PACE), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watson DP, Ray B, Robison L, Xu H, Edwards R, Salyers MP, Hill J, Shue S. Developing Substance Use Programming for Person-Oriented Recovery and Treatment (SUPPORT): protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2017 Dec 15;3:73. doi: 10.1186/s40814-017-0212-1. eCollection 2017. PMID 29270312

RESULTS

PARTICIPANT FLOW:
Groups:
- SUPPORT Group: Subjects enrolled in the intervention.
  SUPPORT clients will be offered 12 months of support service with a recovery coach. The recovery coach will guide the client through their recovery, offering guidance and support, while coordinating their treatment services, including support services. The program will provide clients with up to $700 worth of vouchers to cover the cost of additional flexible support services over the 12 months of program enrollment, which will be personalized to fit the needs of the client. These cost vouchers will cover support services, such as housing, employment services, substance use treatment, transportation, childcare, educational or vocational services, or aftercare planning. The costs of each service is determined by the service provider. Further, the recovery coach will assist the client in choosing appropriate services and coordinating/monitoring service completion.
- Standard Care Group: Subjects enrolled in standard services.
Period: Baseline - 6 Month Follow-Up
Arm/Group | SUPPORT Group | Standard Care Group
Started | 46 | 54
Completed | 19 | 22
Not Completed | 27 | 32
Not completed — Lost to Follow-up | 27 | 32
Period: 6 Month Follow-Up - 12 Month Follow-Up
Arm/Group | SUPPORT Group | Standard Care Group
Started | 19 | 22
Completed | 13 | 20
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUPPORT Group | Standard Care Group | Total
Number analyzed (Participants) | 46 | 54 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 53 | 99
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (8.9) | 38.1 (11.6) | 38.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 26 | 32 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 44 | 53 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 24 | 36
  White | 30 | 30 | 60
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
Sexual Orientation [Count of Participants; unit: Participants]
  Straight | 41 | 51 | 92
  Gay/Lesbian | 3 | 1 | 4
  Bisexual | 1 | 2 | 3
  Other | 0 | 0 | 0
  Don't know/Not Sure | 1 | 0 | 1
Military Status [Count of Participants; unit: Participants]
  Served in military | 1 | 3 | 4
  Not served in military | 45 | 51 | 96
Education Level [Count of Participants; unit: Participants]
  Lower than high school | 9 | 11 | 20
  High school/GED | 21 | 24 | 45
  College or above | 16 | 19 | 35
Housing Status [Count of Participants; unit: Participants]
  Shelter | 8 | 8 | 16
  Street/Outdoors | 2 | 1 | 3
  Institution | 4 | 6 | 10
  Housed: own | 5 | 7 | 12
  Housed: someone else's | 9 | 14 | 23
  Housed: halfway house | 9 | 5 | 14
  Housed: residential treatment | 6 | 12 | 18
  Housed: other | 3 | 1 | 4
Employment Status [Count of Participants; unit: Participants]
  Employed | 6 | 6 | 12
  Unemployed | 40 | 48 | 88
Treatment Motivation [Median (Inter-Quartile Range); unit: score on scale] — The Treatment Motivation Questionnaire (TMQ) is a 26-item instrument. The instrument uses a 7-point scale, ranging from (1) not at all true to (7) very true. The TMQ has four sub scales: internal reasons, external reasons, help seeking, and confidence.
  score on scale
    External Reasons | 2.1 [1.0 to 3.8] | 2.5 [1.3 to 4.0] | 2.4 [1.0 to 3.9]
    Internal Reasons | 6.2 [5.4 to 6.7] | 6.4 [5.5 to 6.8] | 6.3 [5.5 to 6.7]
    Help Seeking | 6.0 [4.8 to 7.0] | 6.5 [5.2 to 7.0] | 6.0 [5.0 to 7.0]
    Confidence | 6.4 [5.2 to 7.0] | 6.6 [5.0 to 7.0] | 6.4 [5.2 to 7.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Substance Use
Description: Using the Frequency of Drug Use scale, we measured self-reported use of alcohol, sedative, tranquilizers, painkillers, stimulants, marijuana, cocaine, crack, hallucinogens, inhalants, heroin, and prescription medications. Respondents are asked to indicate the number of days having used each listed drug within the past 30 days.
  The minimum value is 0, and the maximum value is 30.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 46 | 54
Participants
  0 days alcohol use | 38 | 45
  1-30 days alcohol use | 8 | 9
  0 days illegal drug use | 35 | 43
  1-30 days illegal drug use | 11 | 11
  0 days alcohol or illegal drug use | 32 | 40
  1-30 days alcohol or illegal drug use | 14 | 14

2. Primary Outcome: Number of Participants Reporting Substance Use
Description: as for outcome 1
Time Frame: 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Count of Participants; unit: Participants
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
Participants
  0 days alcohol use | 18 | 14
  1-30 days alcohol use | 1 | 8
  0 days illegal drug use | 17 | 21
  1-30 days illegal drug use | 2 | 1
  0 days alcohol or illegal drug use | 16 | 13
  1-30 days alcohol or illegal drug use | 3 | 9

3. Primary Outcome: Number of Participants Reporting Substance Use
Description: as for outcome 1
Time Frame: 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Count of Participants; unit: Participants
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
Participants
  0 days alcohol use | 13 | 12
  1-30 days alcohol use | 0 | 8
  0 days illegal drug use | 10 | 12
  1-30 days illegal drug use | 3 | 8
  0 days alcohol or illegal drug use | 10 | 12
  1-30 days alcohol or illegal drug use | 3 | 8

4. Primary Outcome: Difference in the Number of Days That Participants Reported Substance Use
Description: as for outcome 1
Time Frame: Baseline- 6 months
Population: Note that analysis was limited to subjects with available data at both time points
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
days
  Number of days using alcohol | 0 [0 to 0] | 0 [0 to 1]
  Number of days using illegal drugs | 0 [0 to 0] | 0 [0 to 0]
  Number of days using alcohol and illegal drugs | 0 [0 to 0] | 0 [0 to 1]

5. Primary Outcome: Difference in the Number of Days That Participants Reported Substance Use
Description: as for outcome 1
Time Frame: 6 months - 12 months
Population: Note that analysis was limited to subjects with available data at both time points
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 10 | 17
days
  Number of days using alcohol | 0 [0 to 0] | 0 [0 to 0]
  Number of days using illegal drugs | 0 [0 to 0] | 0 [0 to 0]
  Number of days using alcohol and illegal drugs | 0 [0 to 0] | 0 [0 to 0]

6. Primary Outcome: Difference in the Number of Days That Participants Reported Substance Use
Description: as for outcome 1
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
days
  Number of days using alcohol | 0 [0 to 0] | 0 [0 to 2]
  Number of days using illegal drugs | 0 [0 to 0] | 0 [0 to 0]
  Number of days using alcohol and illegal drugs | 0 [0 to 0] | 0 [0 to 1.5]

7. Primary Outcome: Difference in Readiness to Change
Description: Stages of Change, Readiness, and Treatment Eagerness Scale (SOCRATES) is a 19-item instrument that measures readiness to change behaviors related to substance use, using a 5 point scale 1 (Strongly Disagree), 2 (Disagree), 3 (Undecided), 4 (Agree), 5 (Strongly Agree). This measure is best used to assess stages of change at baseline; subsequent changes might not be clinically relevant.
  Subscales:
  1. Recognition: A higher score indicates acknowledgement of the problem, possible harm, desires change. (Range: 7-35)
  2. Ambivalence: A higher score reflects openness to reflection on drug use. A lower score may mean they "know" their drug use is causing problems (high Recognition), or they "know" that they do not have drug use problems (low Recognition). Thus, a low Ambivalence score should be interpreted in relation to the Recognition score. (Range: 4-20)
  3. Taking steps: A higher score means steps have been taken, and they may already be experiencing success. (Range: 8-40)
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
score on a scale
  Recognition | -1 [-4 to 0] | -1.08 [-4 to 1]
  Ambivalence | -1 [-4 to 1] | -1 [-3 to 2]
  Taking steps | 0 [-1 to 0] | 0 [-2 to 1]

8. Primary Outcome: Difference in Readiness to Change
Description: as for outcome 7
Time Frame: 6 months - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale
  Recognition | -1 [-7 to 1] | -2 [-9 to 0]
  Ambivalence | -3 [-6 to -0.5] | -1 [-4 to 1]
  Taking steps | 0 [-1 to 2] | 0 [-2 to 0]

9. Primary Outcome: Difference in Readiness to Change
Description: as for outcome 7
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale
  Recognition | -5 [-11 to 0] | -2.5 [-15 to 1]
  Ambivalence | -4 [-8 to -3] | -2 [-5.5 to 0.5]
  Taking steps | 0 [-3 to 4] | -1 [-3.3 to 0.5]

10. Primary Outcome: Difference in Quality of Life: Perceived General Health
Description: Using the 4-item Current Quality of Life Scale, we measured an individual's perceived general physical and mental health during the past 30 days. Self-perception of current physical and mental health is indicative of a person's current health and future health outcomes. The general assessment of health has been shown to be both a solid measure of self-reported health and a powerful predictor of mortality and morbidity.
  One of the four items requests participants to report on their general health, with a scale of (1) excellent, (2) very good, (3) good, (4) fair, (5) poor.
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
score on a scale | 0 [0 to 1] | 0 [-1 to 0]

11. Primary Outcome: Difference in Quality of Life: Perceived General Health
Description: as for outcome 10
Time Frame: 6 months - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale | 0 [-1 to 1] | 0 [-1 to 0]

12. Primary Outcome: Difference in Quality of Life: Perceived General Health
Description: as for outcome 10
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale | 0 [-1 to 0] | 0 [-1 to 0]

13. Primary Outcome: Difference in Quality of Life: Unhealthy Days or Days Limited by Poor Health
Description: Using the 4-item Current Quality of Life Scale, we measured an individual's perceived general physical and mental health during the past 30 days. Self-perception of current physical and mental health is indicative of a person's current health and future health outcomes. The general assessment of health has been shown to be both a solid measure of self-reported health and a powerful predictor of mortality and morbidity.
  Two of the four items requested the number of unhealthy days, physically or mentally, out of the past 30 days. These are reported as a sum.
  One of the four items requested the number of days that usual activities are prevented due to poor physical or mental health are also reported out of the past 30 days.
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
Days
  Number of days physically/mentally unhealthy | -1 [-10 to 9] | 0 [-15 to 0]
  Number of days that usual activities prevented | -2.5 [-7 to 2] | 0 [-13 to 0]

14. Primary Outcome: Difference in Quality of Life: Unhealthy Days or Days Limited by Poor Health
Description: as for outcome 13
Time Frame: 6 months - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
Days
  Number of days physically/mentally unhealthy | -2.5 [-23 to 4] | 0 [-14.5 to 4]
  Number of days that usual activities prevented | 0 [-6 to 1] | 0 [0 to 2.5]

15. Primary Outcome: Difference in Quality of Life: Unhealthy Days or Days Limited by Poor Health
Description: as for outcome 13
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
Days
  Number of days physically/mentally unhealthy | -2 [-30 to 4] | -2 [-16 to 4]
  Number of days that usual activities prevented | -4 [-7 to 0] | 0 [-20 to 0]

16. Primary Outcome: Frequency of Incarceration
Description: Incarceration was measured through publicly available data on arrests, convictions, and periods of incarceration in Indiana. We searched each name in state prison and county jail records and identified them as incarcerated if their name appeared in the jail or prison data during the 12 month study window of their enrollment.
  Note: At baseline, we confirmed with our community partner that each participant had been in prison or jail, or on work release, within the past 3 months. However, this did not match the publicly available data, indicating that the available data is likely incomplete.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 46 | 54
Participants
  Not incarcerated in jail or prison | 28 | 43
  Incarcerated in jail or prison | 18 | 11

17. Primary Outcome: Frequency of Incarceration
Description: as for outcome 16
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 46 | 54
Participants
  Not incarcerated in jail or prison | 30 | 47
  Incarcerated in jail or prison | 16 | 7

18. Secondary Outcome: Difference in Self Determination
Description: The Self-Determination Scale (SDS) assesses individual differences in the extent to which people tend to function in a self-determined way. It is considered a relatively enduring aspect of people's personalities which reflects being more aware of their feelings and sense of self and feeling a sense of choice with respect to their behavior. The SDS is a 10-item scale, with two 5-item subscales: (1) awareness of oneself and (2) perceived choice in one's actions. We utilized only the second scale on perceived choice.
  These 5-items present respondents with 2 statements: Statement (A) indicates more choice and Statement (B) indicates less choice.
  Respondents answer on a five point scale: 1 "Only A feels true", 2 , 3 , 4 , 5 "Only B feels true."
  For perceived choice, the 5 items are reverse scored so that higher scores on every item will indicate a higher level of self-determination. Range: (5-25)
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
score on a scale | 0.2 [-0.4 to 1.2] | 0.3 [-0.4 to 0.8]

19. Secondary Outcome: Difference in Self Determination
Description: as for outcome 18
Time Frame: 6 months - 12 months
Population: Note that analysis was limited to subjects with available data at both time points
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale | 0.2 [0 to 0.4] | 0 [-0.4 to 0.2]

20. Secondary Outcome: Difference in Self Determination
Description: as for outcome 18
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale | 0.7 [-0.2 to 1.2] | 0.5 [0 to 0.8]

21. Secondary Outcome: Difference in Self Efficacy
Description: Using the General Self Efficacy Scale, we measured an individual's belief about whether problems or barriers can be confronted and addressed with a successful outcome. This scale can be used to determine how the respondent copes with daily hassles and adapts to stressful life events. Self-efficacy is indicative of subsequent behavior and can be used for clinical practice and psychological research.
  The 10-item instrument uses a 4-point scale, ranging from 1 (not at all true) to 4 (exactly true), so the composite score ranges from 10 to 40 with higher score indicating greater self-efficacy.
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
score on a scale | 1 [-1 to 3] | 1 [-1 to 5]

22. Secondary Outcome: Difference in Self Efficacy
Description: Using the General Self Efficacy Scale, we measured an individual's belief about whether problems or barriers can be confronted and addressed with a successful outcome. This scale can be used to determine how the respondent copes with daily hassles and adapts to stressful life events. Self-efficacy is indicative of subsequent behavior and can be used for clinical practice and psychological research.
  The 10-item instrument uses a 4-point scale, ranging from 1 (not at all true) to 4 (exactly true), so the composite score ranges from 10 to 40 with higher score indicating greater self-efficacy (a better outcome).
Time Frame: 6 months - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale | -1 [-3 to 1.5] | 1 [-1 to 2]

23. Secondary Outcome: Difference in Self Efficacy
Description: as for outcome 22
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
score on a scale | 4 [-1 to 8] | 1 [-0.5 to 5.5]

24. Secondary Outcome: Difference in Number of Alters That Participants Identified in Their Social Network
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  Respondents identify individuals who make up their social networks. Each individual is identified as an alter, and alters are totaled to determine network size.
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
alters | 0 [-2 to 1] | 0 [-2 to 1]

25. Secondary Outcome: Difference in Number of Alters That Participants Identified in Their Social Network
Description: as for outcome 24
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
alters | 0 [-1 to 0] | 0 [-1 to 2]

26. Secondary Outcome: Difference in the Fraction of Network That Are Close to Subject
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  After identifying their network, respondents are asked to identify how close they are to each alter using a 3-point scale: (1) Very close, (2) Sort of close, (3) Not very close.
  Below is the difference in the fraction of network close to the subject. Results are presented for the fraction of the network identified as being "very close", as well as combined "very close" or "sort of close".
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
alters
  Very close | 0 [-0.07 to 0.25] | 0 [-0.25 to 0.25]
  Very close or sort of close | 0 [0 to 0] | 0 [0 to 0]

27. Secondary Outcome: Difference in the Fraction of Network That Are Close to Subject
Description: as for outcome 26
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
alters
  Very close | 0.33 [-0.08 to 0.57] | -0.07 [-0.25 to 0]
  Very close or sort of close | -0.07 [-0.33 to 0.16] | 0 [-0.03 to 0.0]

28. Secondary Outcome: Difference in the Network Closeness Sum
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  Network closeness refers to the closeness of the participant's network (i.e. how close the alters identified are to one another).
  After identifying alters within their network, respondents are asked to identify how close each alter is to one another using a 3-point scale: (1) Very close, (2) Sort of close, (3) Not very close. Thus, for each original alter pair, the respondent scores their closeness on a range of 1 to 3. A lower score indicates a stronger network.
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 16 | 20
score on a scale | -0.5 [-5.5 to 1] | -1 [-5 to 2]

29. Secondary Outcome: Difference in the Network Closeness Sum
Description: as for outcome 28
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 9 | 18
score on a scale | 0.5 [-1.5 to 3] | 0.5 [-5 to 5]

30. Secondary Outcome: Difference in the Network Closeness Average
Description: as for outcome 28
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 16 | 20
score on a scale | 0 [-0.25 to 0.3] | 0.17 [-0.33 to 0.58]

31. Secondary Outcome: Difference in the Network Closeness Average
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters. This component focuses on the closeness of the participants network (i.e. how close the alters identified are to one another).
  After identifying alters within their network, respondents are asked to identify how close each alter is to one another using a 3-point scale: (1) Very close, (2) Sort of close, (3) Not very close. Thus, for each alter pair, the respondent scores their closeness on a range of 1 to 3, with a lower score indicating more closeness.
  Below is the difference in the network closeness. The range for this scale will differ, depending on the number of alters identified.
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 9 | 18
score on a scale | 0.37 [-0.5 to 0.83] | 0.33 [-0.33 to 0.4]

32. Secondary Outcome: Difference in the Network Closeness Density
Description: as for outcome 28
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 16 | 20
score on a scale | 0.18 [0 to 0.42] | 0 [0 to 0.4]

33. Secondary Outcome: Difference in the Network Closeness Density
Description: as for outcome 28
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 9 | 18
score on a scale | 0.08 [-0.07 to 0.42] | 0 [0 to 0.1]

34. Secondary Outcome: Difference in the Fraction of Network Communicating With Subject
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  After identifying their network, respondents are asked to identify how often they see this person or talk to them on the phone or video chat using a 3-point scale (1) Often, (2) Occasionally, (3) Hardly Ever. Below is the difference in the fraction of network communicating with the subject. Results are presented for the fraction of the network identified as communicating "often", as well as combined "often" or "occasionally".
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
alters
  Often | 0 [0 to 0.25] | 0 [-0.25 to 0.08]
  Often or occasionally | 0 [0 to 0] | 0 [0 to 0]

35. Secondary Outcome: Difference in the Fraction of Network Communicating With Subject
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  After identifying their network, respondents are asked to identify how often they see this person or talk to them on the phone or video chat using a 3-point scale(1) Often, (2) Occasionally, (3) Hardly Ever. Below is the difference in the fraction of network communicating with the subject. Results are presented for the fraction of the network identified as communicating "often", as well as combined "often" or "occasionally".
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
alters
  Often | 0.17 [0 to 0.40] | 0 [-0.25 to 0.09]
  Often or occasionally | 0 [-0.15 to 0] | 0 [0 to 0]

36. Secondary Outcome: Difference in the Fraction of Network Providing Support to the Subject
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  After identifying their network, respondents are asked to identify types of support provided by alters. Examples are given (listed below) and subjects select all that apply. Below is the difference in the fraction network providing support to the subject.
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
alters
  Listens when they are feeling down or upset | 0 [0 to 0.25] | 0 [0 to 0]
  Tells them they care about what happens to them | 0 [0 to 0] | 0 [-0.17 to 0]
  Gives suggestions to them when they have a problem | 0 [0 to 0.25] | 0 [0 to 0.20]
  Tries to help them with daily chores | 0 [-0.14 to 0.25] | 0 [-0.04 to 0.50]
  Helps them out when they are short on money | 0 [0 to 0.42] | 0 [-0.47 to 0.25]

37. Secondary Outcome: Difference in the Fraction of Network Providing Support to the Subject
Description: as for outcome 36
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
alters
  Listens when they are feeling down or upset | 0 [0 to 0.33] | 0 [0 to 0]
  Tells them they care about what happens to them | 0 [-0.17 to 0] | 0 [0 to 0]
  Gives suggestions to them when they have a problem | 0.19 [0 to 0.25] | 0 [0 to 0]
  Tries to help them with daily chores | 0 [-0.17 to 0.23] | 0 [-0.33 to 0.33]
  Helps them out when they are short on money | 0.21 [0 to 0.43] | 0 [-0.25 to 0.17]

38. Secondary Outcome: Difference in the Fraction of Network Causing Subject Problems
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  After identifying their network, respondents are asked to identify whether the alter ever hassles them, causes them problems, or makes life difficult, using a 3-point scale: (1) A lot, (2) Sometimes, (3) No/Not Really. Below is the difference in the fraction of network causing the subject problems. For analysis, we combined "a lot" and "sometimes" into a single category and compared it to "no/not really".
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
alters | 0 [-0.33 to 0.14] | 0 [-0.14 to 0.25]

39. Secondary Outcome: Difference in the Fraction of Network Causing Subject Problems
Description: as for outcome 38
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
alters | -0.29 [-0.50 to 0.14] | 0 [-0.25 to 0]

40. Secondary Outcome: Difference in the Fraction of Network Using Substance(s)
Description: The Social Networks tool is an interviewer-administered questionnaire to assess whom respondents depend on for help in important general matters and specific health matters. This measure captures each of the respondent's network members and a complete assessment of network structure to construct the respondent's social network and whom they rely on for help with health-related and other matters.
  After identifying their network, respondents are asked to identify whether the alter uses alcohol, tobacco, or illicit drugs/medication for reasons other their prescribed purposes. Below is the difference in the fraction of the network using a substance(s).
Time Frame: Baseline - 6 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 19 | 22
alters
  Alcohol | 0 [-0.33 to 0.25] | 0 [-0.09 to 0.16]
  Tobacco | 0 [0 to 0.17] | -0.07 [-0.27 to 0]
  Drugs | 0 [0 to 0] | 0 [-0.17 to 0]

41. Secondary Outcome: Difference in the Fraction of Network Using Substance(s)
Description: as for outcome 40
Time Frame: Baseline - 12 months
Population: Note that analysis was limited to subjects with available data at both time points.
Measure: Median (Inter-Quartile Range); unit: alters
Arm/Group | SUPPORT Group | Standard Care Group
Number analyzed (Participants) | 13 | 20
alters
  Alcohol | -0.04 [-0.33 to 0] | 0 [-0.17 to 0.21]
  Tobacco | 0 [-0.27 to 0.08] | -0.19 [-0.33 to 0]
  Drugs | 0 [-0.08 to 0.14] | 0 [-0.15 to 0]

ADVERSE EVENTS:
Time Frame: Each SUPPORT participant was enrolled in the study for 15 months, and each standard care participant was enrolled in the study for 12 months. Adverse event data was collected for the duration of study enrollment.
Arm/Group | SUPPORT Group | Standard Care Group
All-Cause Mortality (participants affected / at risk) | 2/46 | 1/54
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/54
Other Adverse Events (participants affected / at risk) | 0/46 | 0/54

LIMITATIONS AND CAVEATS:
A limitation is that this is a pilot study for which formal hypothesis testing was not a goal. Retention was low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03132753/Prot_SAP_001.pdf
  • Informed Consent Form (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT03132753/ICF_000.pdf